CLINICAL TRIAL: NCT00623675
Title: Heavy Metal Urine Analysis in 20 Healthy Persons Taking Mineralox
Status: Suspended | Phase: Phase 4 | Type: Interventional
Sponsor: CreoMed, Inc. (Industry)
Responsible Party: Joseph Pergolizzi, Jr., MD, NEMA Research, Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZEO-002
Record Dates: First submitted 2008-02-17; First posted 2008-02-26 (Estimated); Last update posted 2009-07-07 (Estimated); Status verified 2009-07

CONDITIONS: Healthy
Keywords: zeolites; nutraceuticals; natural supplements; Healthy volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Dietary Supplement: Mineralox C

INTERVENTIONS:
Dietary Supplement: Mineralox C — Mineralox C 2 capsules three times a day.

SUMMARY:
Researchers want to find out if urine heavy metal levels are changed in persons who use Mineralox Basic C™ (Mineralox). Mineralox is a zeolite (clinoptilolite) in combination with Vitamin C. Zeolites are natural supplements (nutraceuticals) that work at the cellular level to remove heavy metals and toxins that are accumulated in every day life safely from the body through the urine. The study doctor will give Mineralox to 20 people in this study to see if it helps with the heavy metal removal from the body.

ELIGIBILITY:
Inclusion Criteria:

1. Females and Males age 18-75 without significant health problems as determined by the Principal Investigator.
2. Nonsmoker
3. Ability to understand informed consent

Exclusion Criteria:

1. Pregnancy
2. Any serious or unstable disease within 6 months; seizure risk; diabetes mellitus requiring insulin or oral hypoglycemic medication; diagnosis of eating disorder, use of MAOI in the prior 14 days; hepatic or renal impairment; clinically significant cardiovascular disease within 6 months; uncontrolled hypertension; severe chronic obstructive pulmonary disease; baseline systolic blood pressure higher than150mm Hg or diastolic blood pressure higher than 95 mm Hg; history of cancer (except treated basal cell or squamous cell carcinoma of the skin); history of clinically significant allergic reactions or laboratory abnormalities,and patients taking AREDS Eye Vitamins.
3. Major depressive disorder within the past year requiring treatment; history of panic disorder, psychosis, bipolar disorder, or eating disorder
4. Intention to donate blood or blood products during treatment phase of the study;
5. Alcohol or drug abuse/dependency within the past year
6. Use of tobacco products other than cigarettes or use of marijuana
7. Body mass index (calculated as weight in kilograms divided by the square height in meters) less than 15 or greater than 38 or weight less than 45.5 kg
8. NRT, antidepressants, antipsychotics, mood stabilizers/anticonvulsants, naltrexone, steroids or insulin.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-02

PRIMARY OUTCOMES:
Heavy Metal Urine Analysis | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Joseph V Pergolizzi, MD, Principal Investigator — NEMA Research, Inc.
Locations (1):
- NEMA Research, Naples, Florida, United States